CLINICAL TRIAL: NCT05853094
Title: A Single-centre, Randomized Study to Compare the Outcomes of Protected Transverse Colostomy Versus Ileostomy After Low Anterior Resection of Low Rectal Cancer From the Perspective of Intestinal Microecology
Brief Title: Postoperative Effects of Different Enterostomy Approaches
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Ma Yanlei, Chief Physician, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDCRC88-MYL
Record Dates: First submitted 2023-04-10; First posted 2023-05-10 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms Malignant; Intestinal Neoplasms, Malignant
Keywords: Colorectal Cancer; Stoma
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Intestinal Neoplasms | interventions — Ileostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ileostomy (Experimental): Protective ileostomy as a defunction mean after low anterior resection
  Interventions: Procedure: Ileostomy
- Transverse colostomy (Experimental): Protective transverse colostomy as a defunction mean after low anterior resection
  Interventions: Procedure: Transverse colostomy

INTERVENTIONS:
Procedure: Ileostomy — Protective loop ileostomy after low anterior resection
  Arms: Ileostomy
Procedure: Transverse colostomy — Protective loop transverse colostomy after low anterior resection
  Arms: Transverse colostomy

SUMMARY:
Exploring the effect of protective ileostomy compared with transverse colostomy on the occurrence of complications, the occurrence of serious side effects of adjuvant chemotherapy and disease recurrence in patients with low rectal cancer after radical surgery from the perspective of intestinal microecology.

DETAILED DESCRIPTION:
Low rectum refers to the rectal area <7 cm from the anal verge. At present, with the development of modern medical technology and the change of surgical concept, more and more patients can achieve the goal of radical treatment of low rectal cancer while preserving the anus. The occurrence of anastomotic leakage after anus-preserving surgery for low-grade rectal cancer is a more common and serious complication, with an incidence ranging from 2.4% to 15.9%, and the morbidity and mortality rate after anastomotic leakage can be as high as 16%.

A protective stoma protects the anastomosis by temporarily establishing an artificial channel above the anastomosis to divert feces and avoid mechanical pressure and contamination of the anastomosis by intestinal contents, allowing the anastomosis to grow and heal in relatively clean external conditions. The current choices of protective stoma sites are terminal ileum and transverse colon. Analysis of domestic and international studies shows that both protective transverse colostomy and ileostomy can achieve the effect of diversion of stool, but whether there is a difference in preventing anastomotic leakage and reducing adverse outcomes of anastomotic leakage remains to be investigated. There are significant inconsistencies between domestic and international studies regarding the incidence of stoma-related complications caused by different stoma sites: the study by Rondelli et al. showed that terminal ileostomy was associated with lower stoma-related complications, and a domestic meta-analysis recommended terminal ileostomy after radical rectal cancer surgery. In contrast, the study by the team from the Union Hospital showed that transverse colostomy was associated with significantly lower rates of stoma-related complications and perioperative complications of stoma reentry.

In addition, according to the Union Hospital team study, the incidence of postoperative intestinal microbiota dysbiosis was higher in patients who underwent ileostomy compared to those who underwent transverse colostomy. The total intestinal microbiota in the colon accounts for more than 90% of the systemic intestinal microbiota, and the intestinal microbiota in the large intestine can be roughly restored to preoperative levels after transverse colostomy, whereas a large amount of intestinal microbiota is lost and difficult to restore after ileostomy. The dominant flora in the colon, such as Clostridium and Enterococcus, are less likely to colonize the small intestine, which may adversely affect the intestinal and systemic immune regulation and antitumor immune effects of the body. In addition, patients with progressive low-grade rectal cancer routinely require adjuvant chemotherapy after radical surgery, and there are no studies at domestic or abroad on whether terminal ileostomy, which is more common than transverse colostomy for intestinal dysbiosis, has any differences on the efficacy and toxic side effects of adjuvant chemotherapy for patients; furthermore, it is also important to investigate whether the two different stoma methods have an impact on long-term disease recurrence and overall survival of patients. In addition, whether the two different stoma modalities have an effect on long-term disease recurrence and overall survival is also an important research question.

Therefore, the investigators propose to conduct a prospective, randomized, controlled study in patients with low-grade rectal cancer who underwent radical surgery (with or without neoadjuvant radiotherapy) to investigate whether there are differences in the incidence of complications, serious side effects of adjuvant chemotherapy, and disease recurrence after terminal ileostomy versus transverse colostomy from the perspective of intestinal microecology, and to explore the differences in systemic immunity, inflammatory, and metabolic status.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological confirmed adenocarcinoma of the rectum;
2. Patients age between 18-80;
3. Baseline AJCC stage I-III: cT1-4N0-2M0 (AJCC-8 version);
4. Eastern Cooperative Oncology Group (ECOG) physical status score of 0 to 2;
5. Patients voluntarily sign informed consent.

Exclusion Criteria:

1. Other types of rectal cancer (adenosquamous carcinoma, squamous carcinoma, neuroendocrine tumors, clear cell carcinoma, spindle cell carcinoma, undifferentiated carcinoma);
2. Combination of rectal cancer with multiple carcinomas;
3. Pre-operative presence of acute and chronic infectious diseases or foci of infection;
4. Intraoperative radical surgery was not performed for various reasons；
5. Colostomy was not performed at the same time as the radical rectal cancer surgery;
6. Combined with intestinal obstruction, intestinal perforation, intestinal bleeding, peritonitis, etc. requiring emergency surgery;
7. Metastatic cancer;
8. Serious heart, lung, liver and kidney disease, can not tolerate surgery;
9. Active liver disease or abnormal liver function with ALT, AST and TBIL more than 2 times the upper limit of normal values;
10. Renal impairment with Cr ≥ 2 times the upper limit of normal or BUN ≥ 2 times the upper limit of normal;
11. Blood leukocytes below the lower limit of normal value, or platelets below the lower limit of normal value, or with other blood system diseases;
12. Pregnancy;
13. Mental illness or serious intellectual disability who cannot describe their feelings correctly;
14. Severe coagulation disorder, bleeding tendency;
15. Patients with severe uncontrolled medical disease, recent history of myocardial infarction (within 3 months), uncontrolled severe hypertension and severe diabetes mellitus;
16. Patients need to be on antibiotics/other probiotics for a long time.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-06-23 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Microbiome functional gene capacity in postoperative stoma pouch and distal intestine by metagenomic sequencing | 1 month
  Determining the structural impact of different stoma methods on intestinal microecology by metagenomic sequencing
Microbiome functional gene capacity in postoperative stoma pouch and distal intestine by metagenomic sequencing | 6 months
  Determining the structural impact of different stoma methods on intestinal microecology by metagenomic sequencing
Microbiome functional gene capacity in postoperative stoma pouch and distal intestine by metagenomic sequencing | 3 years
  Determining the structural impact of different stoma methods on intestinal microecology by metagenomic sequencing

SECONDARY OUTCOMES:
Concentration of inflammatory markers | 1 month
  Measurement of plasma inflammatory markers such as IL-6, TNF-α, CRP and PCT
Changes in cellular immunity status | 1 month
  Estimation of dynamics of cellular immunity as measured by the proportion of CD3+, CD4+, CD8+, CD4+CD25+CD127low, CD16+CD56+ cells using flowcytometry
Changes in humoral immunity status | 1 month
  Estimation of dynamics of humoral immunity as measured by the proportion of CD3-CD19+, CD20+ cells using flowcytometry
Incidence of anastomotic leakage | 1 month
  The occurrence of postoperative anastomotic leakage
Early postoperative complications rate | 1 month
  Incidence of postoperative complications such as diarrhea, intestinal obstruction, incisional infection, stoma prolapse, stoma necrosis, parastomal hernia, irritant dermatitis, renal insufficiency, etc.
First intestinal gas time | 1 month
  Documenting the patient's post-operative recovery
First defecation time | 1 month
  Documenting the patient's post-operative recovery
Concentration of inflammatory markers | 6 month
  Measurement of plasma inflammatory markers such as IL-6, TNF-α, CRP and PCT
Changes in cellular immunity status | 6 month
  Estimation of dynamics of cellular immunity as measured by the proportion of CD3+, CD4+, CD8+, CD4+CD25+CD127low, CD16+CD56+ cells using flowcytometry
Changes in humoral immunity status | 6 month
  Estimation of dynamics of humoral immunity as measured by the proportion of CD3-CD19+, CD20+ cells using flowcytometry
Incidence of grade 3-4 serious side effects of adjuvant chemotherapy | 6 month
  Assessed with Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Adjuvant chemotherapy toxicity and quality of life scores | 6 months
  Assessed with European Organization for Research and Treatment of Cancer high-dose chemotherapy specific quality of life questionnaire module (EORTC QLQ-HDC29), ranging from 29 to 116 and higher scores suggest worse quality of life
Concentration of inflammatory markers | 3 years
  Measurement of plasma inflammatory markers such as IL-6, TNF-α, CRP and PCT
Changes in cellular immunity status | 3 years
  Estimation of dynamics of cellular immunity as measured by the proportion of CD3+, CD4+, CD8+, CD4+CD25+CD127low, CD16+CD56+ cells using flowcytometry
Changes in humoral immunity status | 3 years
  Estimation of dynamics of humoral immunity as measured by the proportion of CD3-CD19+, CD20+ cells using flowcytometry
Disease-free Survival | 3 years
  Time between the start of surgical randomization and recurrence of disease or death (from any cause)Time between the start of surgical randomization and recurrence of disease or death (from any cause)
Overall Survival | 3 years
  Time from the start of surgical randomization to death (from any cause)

CONTACTS AND LOCATIONS:
Overall Officials: Yanlei Ma, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China